CLINICAL TRIAL: NCT01166568
Title: A Prospective, Multicenter Clinical Trial Of the PresVIEW Scleral Implant (PSI) For the Improvement Of Near Visual Acuity In Presbyopic Patients
Brief Title: Trial of the PresVIEW Implant for the Improvement of Near Vision in Patients With Presbyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Refocus Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-277-5
Record Dates: First submitted 2010-07-16; First posted 2010-07-21 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Presbyopia
Keywords: Presbyopia; Reading Vision; Near Vision
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Intervention Model Description: A non-randomized arm was run in parallel with a randomized sub-study consisting of 2 arms; Immediate Treatment and Deferred Treatment. Upon completion of the 6 month observation period, the Deferred Treatment group then crosses over upon implantation to become part of the overall study group.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Implantation-Non Randomized (Experimental): Subjects are not participants in the randomized sub-study. PresView Scleral Implants surgical placed in the eye(s) after enrollment and meeting inclusion/exclusion criteria.
  Interventions: Device: PresVIEW Scleral Implants
- Implantation-Randomized (Experimental): Subjects are participants in the randomized sub-study. Subjects were randomized to the Immediate Treatment group. PresView Scleral Implants surgical placed in the eye(s)Subjects are participants in the randomized sub-study after enrollment and meeting inclusion/exclusion criteria.
  Interventions: Device: PresVIEW Scleral Implants
- Deferred Implantation-Randomized (No Intervention): Subjects are participants in the randomized sub-study after enrollment and meeting inclusion/exclusion criteria. Subjects were randomized to the Deferred Treatment group are observed for 6 months. Upon completion of the observation follow-up, subjects can opt to have PresView Scleral Implants surgically placed in the eye(s) and become part of the overall study experimental group.

INTERVENTIONS:
Device: PresVIEW Scleral Implants — Subjects are implanted with the PresView Scleral Spacing Implants and followed for 24 months.
  Arms: Implantation-Non Randomized; Implantation-Randomized

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of the PresVIEW™ Scleral Implant (PSI) for the improvement of near visual acuity in presbyopic patients.

DETAILED DESCRIPTION:
The clinical investigation of the PresView™ Scleral Implant (PSI) is a prospective multicenter clinical trial in which a total of 330 subjects were enrolled and implanted with the PSI and followed for a period of 24 months at up to 14 clinical sites.

An additional randomized sub-study was performed on 48 subjects with the PSI Second Generation PresView™(SGP) implant, model number SGP-046. A 2:1 randomization was used to determine the 32 subjects assigned to be implanted and the 16 subjects assigned to the observation/deferred implantation control arm. Subjects randomized to the deferred implantation control arm were eligible to receive the PSI after completion of the 6 months of observation in the study.

All subjects interested in participating in the study were screened for eligibility, and informed consent was obtained from those who meet the inclusion/exclusion criteria. Eligible subjects were examined preoperatively to obtain a medical history and baseline ocular data.

Effectiveness: The following tests/measurements used to evaluate the effectiveness of the PSI procedure will be included in the study protocol:

* Near visual acuity of the operated eye/eyes as compared with baseline (uncorrected and distance corrected)
* Reading acuity of the operated eye/eyes as compared with baseline (uncorrected and distance corrected)

The PSI procedure will be defined as successful if a logMar equivalent to Snellen 20/40 or better (logMar 0.3) is achieved in ≥ 75% of patients or if 75% of patients realize an improvement ≥ 2 lines in distance corrected near visual acuity (DCNVA). For most patients, this will translate into the ability to read the majority of newspaper and magazine print without a near optical aid.

Safety: Primary safety outcomes for safety will include:

* Incidence of anterior segment ischemia
* Decrease in Best Corrected Distance Visual Acuity (BCDVA) of more than 2 lines from baseline at 1-month or more postoperatively
* Decrease in best distance corrected near acuity (with add) of more than 2 lines from baseline at 1-month or more postoperatively
* Intraocular Pressure (IOP) increase > 10mm Hg over baseline or IOP > 25mm Hg after 1 Day postoperative
* Signs of chronic inflammation (e.g. uveitis or chronic conjunctival hyperemia) at 2 months or more postoperatively
* Increase in axial length of ≥ 0.20mm accompanied by a > 0.5 diopter myopic shift in manifest spherical equivalent distance refraction.
* Incidence of adverse events: total not to exceed 5%, and the incidence of each event should not exceed 1-2%

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 50-60 years old
* Subject must have a best corrected distance visual acuity of 20/20 or better
* Subject must have SLOAN distance corrected near visual acuity @ 40cm in the operative eye/eyes of 20/50 to 20/100 (inclusive).
* Subject should have a manifest distance spherical equivalent refractive correction in the operative eye/eyes of from -0.50 to +0.75 diopters with no more than 1.00 diopter of astigmatism and should require at least a +1.50 diopter add. The distance manifest refraction spherical equivalent and the distance cycloplegic refraction spherical equivalent must be within 0.50 diopters of each other.
* Subject must be phakic in the study eye
* Subject must be mentally competent to understand and comply with the requirements of the study.
* Subject must be able to provide written informed consent.

Exclusion Criteria:

* Chronic uveitis or other recurrent anterior or posterior segment inflammation in either eye.
* Scleral thickness less than 530 μm in the operative eye/eyes.
* Any previous eye surgeries including cataract, LASIK, or Muscle surgery
* Any history of prior extraocular muscle surgery, specifically the recti or oblique muscles.
* Any chronic systemic diseases such as diabetes, heart disease, Lupus, etc.
* Any eye diseases such as eye inflammation, infection, cataract, or retinal diseases
* Allergic to any medications used in the study.
* The patient may not have participated in a device clinical study for the operative eye within the last 3 months and may not have been implanted with PSI devices in this or any other study.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 337 (Actual)
Dates: Start 2003-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schanzlin, M.D., Principal Investigator — Chief Medical Officer
Locations (14):
- United States (14):
  - Boxer-Wachler Vision Institute, Beverly Hills, California
  - Gordon-Weiss-Schanzlin Vision Institute, San Diego, California
  - The Midwest Center for Sight, Des Plaines, Illinois
  - Jacksoneye, Lake Villa, Illinois
  - Vision/Advanced Eye Center, Lombard, Illinois
  - The Eye Care Institute, Louisville, Kentucky
  - Associated Vision Consultants, Southfield, Michigan
  - Cornea Associates, Omaha, Nebraska
  - Fichte, Endl and Elmer Eyecare Creekside Center, Amherst, New York
  - Southeastern Eye Center, Greensboro, North Carolina
  - Eye Associates of South Tulsa, Tulsa, Oklahoma
  - Wang Vision Institute, Nashville, Tennessee
  - Braverman-Terry-Oei-Eye Associates, San Antonio, Texas
  - The Center for Corrective Eye Surgery, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: US Food and Drug Administration Website — http://www.fda.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The prospective, multicenter clinical trial of the PresView Implant was conducted at 14 clinical sites. All recruitment evaluations were performed at the Principal Investigator's sites and subjects were screened for eligibility. If inclusion/exclusion criteria were met, informed consent was obtained and the subject was enrolled in the study.
Pre-assignment Details: Once determined eligible and informed consent was obtained, both eyes were enrolled in the study. Per protocol, primary outcome analysis must be performed on the primary eye only and the primary eye is therefore the unit of analysis. Fellow eyes were followed for safety outcomes and summarized separately.
Units Other Than Participants: Eye
Groups:
- PresVIEW Implantation - Non-Randomized: Subjects in the non-randomized arm of the study were bilaterally implanted and followed for 24 months. Per the protocol, primary endpoint analysis was performed on the primary eye (only). Fellow eyes were followed for safety and summarized separately
- PresVIEW Implantation - Randomized: A randomized sub-study was used to evaluate the early (6 Month) effectiveness of the PresVIEW™ Scleral Implants against a deferred control group (no treatment). Subjects in the randomized sub-study that were randomly assigned to the immediate treatment (surgical) group were bilaterally implanted and followed for 24 months. Pre-operative, 3 month and 6 month post-operative visual acuity for the primary eye was compared to the differed treatment group primary eye visual acuity results. Thirty-two subjects of the total 48 subjects participating in the randomized sub-study, were randomly assigned to receive immediate surgery.
- PresVIEW Deferred Implantation - Randomized: Subjects in the randomized sub-study that were randomly assigned to the deferred treatment (control) group were bilaterally implanted after 6 months observation and followed for 24 months post-op. Sixteen subjects of the total 48 subjects participating in the randomized sub-study were randomly assigned to the control group and followed for 6 months prior to surgery (observation). These patients will provide additional informed consent for implantation and their results will be included in the total patient cohort for the PSI SGP-046. Total study participation will be either 6 months (if they did not elect treatment after 6 months observation), or 30 months (6 months observation + 24 months post-operative) if they elected treatment. The observation period included follow-up visits for Day 0 (baseline), 3 months, and 6 months for the randomized sub-study and visual acuity for the primary eye was compared to the immediate treatment group primary eye visual acuity for analysis.
Period: Deferred Implantation- Randomized
Arm/Group | PresVIEW Implantation - Non-Randomized | PresVIEW Implantation - Randomized | PresVIEW Deferred Implantation - Randomized
Started | 0; 0 Eye | 0; 0 Eye | 16; 32 Eye
Completed | 0; 0 Eye | 0; 0 Eye | 15; 30 Eye (From the randomized sub-study control group (n=16), 1 subject withdrew during the observation phase)
Not Completed | 0; 0 Eye | 0; 0 Eye | 1; 2 Eye
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Implantation- Nonrandomized & Randomized
Arm/Group | PresVIEW Implantation - Non-Randomized | PresVIEW Implantation - Randomized | PresVIEW Deferred Implantation - Randomized
Started | 288; 562 Eye | 33; 66 Eye | 9; 17 Eye (15 subjects completed the observation phase and 9 subjects (17 eyes) proceeded with implantation.)
Completed | 274; 537 Eye | 32; 64 Eye | 8; 16 Eye ((1) Primary eye implanted only subject withdrew consent after implantation of the device.)
Not Completed | 14; 25 Eye | 1; 2 Eye | 1; 1 Eye
Not completed — Lost to Follow-up | 7 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Between 50 to 60 years of age at the commencement of the study.
Groups:
- PresVIEW Implantation Non-Randomized: 288 subjects that received the PresView Scleral Implants, which were surgical placed in the sclera of the eye. Subjects were followed for 24 months. This sample consists of; 16 randomized deferred implantation subjects, 32 randomized implantation subjects, and 282 non-randomized implanted subjects (i.e. all enrolled subjects).
- PresVIEW Implantation - Randomized: 33 randomized subjects entered into a immediate treatment (implantation) group. Subjects were followed for 24 months. Immediate treatment group data was compared to the Deferred Treatment group at 6 months.
- PresVIEW Deferred Implantation - Randomized: 16 randomized subjects entered into a deferred treatment (control) group arm. Subjects were followed for 6 months (observation). Subjects that completed the 6 month observation were then offered PresVIEW implantation.
- Total: Total of all reporting groups
Arm/Group | PresVIEW Implantation Non-Randomized | PresVIEW Implantation - Randomized | PresVIEW Deferred Implantation - Randomized | Total
Number analyzed (Participants) | 288 | 33 | 16 | 337
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.92 (2.90) | 54.62 (2.96) | 55.03 (2.66) | 54.93 (2.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 15 | 8 | 151
  Male | 160 | 18 | 8 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 6 | 2 | 40
  Not Hispanic or Latino | 256 | 27 | 14 | 297
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 0 | 4
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 0 | 0 | 12
  White | 258 | 27 | 14 | 299
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 6 | 2 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 288 | 33 | 16 | 337
DCNVA 20/40 or Better (at baseline) [Count of Participants; unit: Participants] | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Primary Eyes With Distance Corrected Near Visual Acuity (DCNVA) to 20/40 or Better or Improvement of 2 or More Lines
Description: Measurement of the Distance Corrected Near Visual Acuity at 40 centimeters achieving 20/40 or better or improvement of 2 or more lines at 24 months for the primary eye.
Time Frame: From date of baseline measurement until the date of study withdrawal or study completion, whichever came first, assessed up to 2 years.
Population: Explanted primary eyes were analyzed as failures. Data for primary eyes that missed the 24 month visit, were lost to follow-up, or withdrew consent prior to the 24 month visit were not imputed. Per protocol, primary outcome analysis must be performed on the primary eye only. Fellow eye data is used for safety outcomes and summarized separately.
Measure: Count of Units; unit: Primary Eyes
Units Other Than Participants: Primary Eyes
Groups:
- Overall Study Population: A total of 330 subjects at 11 sites received implantation of the PSI and were followed for 24 months post surgical. As per the protocol, the primary eye is the unit of analysis and was used for primary endpoint analysis. Fellow eyes were followed for safety and summarized separately. The primary eyes of subjects participating in the randomized sub-study were analyzed separately, though, they were also considered part of the overall study if they received implantation of the PSI.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 317
Number analyzed (Primary Eyes) | 317
Primary Eyes | 288
Statistical Analysis 1: Comparison: Overall Study Population; The PSI procedure is defined as successful if 75% of subjects achieve the first primary endpoint or second primary endpoint. The corresponding statistical hypotheses are as follows: H0 (null hypothesis): p1 ≤ 0.75 Ha (alternative hypothesis): p1 > 0.75, Where, p1 is the probability of subjects achieving the first primary endpoint. H0 (null hypothesis): p2 ≤ 0.75 Ha (alternative hypothesis): p2 > 0.75, Where, p2 is the probability of subjects achieving the second primary endpoint; Test type: Superiority; p = 0.025, Fisher Exact — the p-value is adjusted for multiple comparisons; binomial distribution = 0.75, 97.5% CI 1-sided [lower limit 0.75]

2. Secondary Outcome: Presence of Significant Safety Events (SAEs).
Description: The point estimate were calculated for clinically significant adverse events (SAE's) at the end of the study. Incidence of adverse event totals should not to exceed 5%, and the incidence of each event should not exceed 1-2%.
  NOTE: Because the secondary outcome is a safety measure, both primary and fellow eyes were used for analysis.
Time Frame: From initiation of the implantation procedure (operative day) until study completion at 24 months or withdrawal from the study.
Population: All subject eyes implanted with the PSI were included in the safety analysis. The point estimates were calculated for each of the following events at 24 months. Only the incidence of serious adverse events (SAE's) is presented here as only (1) secondary outcome is allowed.
Measure: Count of Units; unit: Primary and Fellow Eyes
Units Other Than Participants: Primary and Fellow Eyes
Groups:
- Overall Study Population: A total of 330 subjects at 11 sites received implantation of the PSI and were followed for 24 months post surgical. For the safety analysis, subjects participating in the randomized sub-study were analyzed as part of the overall study if they received implantation of the PSI.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 330
Number analyzed (Primary and Fellow Eyes) | 645
Primary and Fellow Eyes | 3

3. Other Pre Specified Outcome: Safety Parameter Point Estimate -- Anterior Segment Ischemia
Description: All primary and fellow eyes implanted with the PSI were included in the safety analysis. Point estimates were calculated for the incidence of Anterior Segment Ischemia at the end of the study. Incidence of adverse event totals should not to exceed 5%, and the incidence of each event should not exceed 1-2% NOTE: Because the secondary outcome is a safety measure, both primary and fellow eyes were used for analysis.
Time Frame: as for outcome 2
Population: All subject eyes implanted with the PSI were included in the safety analysis.
Measure: Count of Units; unit: Primary and Fellow Eyes
Units Other Than Participants: Primary and Fellow Eyes
Groups:
- Overall Study Population: A total of 330 subjects (645 eyes) at 11 sites received implantation of the PSI and were followed for 24 months post surgical. For the safety analysis, subjects participating in the randomized sub-study were analyzed as part of the overall study if they received implantation of the PSI.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 330
Number analyzed (Primary and Fellow Eyes) | 645
Primary and Fellow Eyes | 0

4. Other Pre Specified Outcome: Safety Parameter Point Estimate -- Decrease in BCDVA > 2 Lines
Description: All primary and fellow eyes implanted with the PSI were included in the safety analysis. Point estimates were calculated for the incidence of Decrease in BCDVA > 2 lines at the end of the study. Incidence of adverse event totals should not to exceed 5%, and the incidence of each event should not exceed 1-2%.
  NOTE: Because the secondary outcome is a safety measure, both primary and fellow eyes were used for analysis.
Time Frame: as for outcome 2
Population: All subject eyes implanted with the PSI were included in the safety analysis.
Measure: Count of Units; unit: Primary and Fellow Eyes
Units Other Than Participants: Primary and Fellow Eyes
Arm/Group | Overall Study Population
Number analyzed (Participants) | 330
Number analyzed (Primary and Fellow Eyes) | 645
Primary and Fellow Eyes | 1

5. Other Pre Specified Outcome: Safety Parameter Point Estimate -- Decrease in BCNVA > 2 Lines
Description: All primary and fellow eyes implanted with the PSI were included in the safety analysis. Point estimates were calculated for the incidence of Decrease in BCNVA > 2 lines at the end of the study. Incidence of adverse event totals should not to exceed 5%, and the incidence of each event should not exceed 1-2%.
  NOTE: Because the secondary outcome is a safety measure, both primary and fellow eyes were used for analysis.
Time Frame: as for outcome 2
Population: All subject eyes implanted with the PSI were included in the safety analysis.
Measure: Count of Units; unit: Primary and Fellow Eyes
Units Other Than Participants: Primary and Fellow Eyes
Arm/Group | Overall Study Population
Number analyzed (Participants) | 330
Number analyzed (Primary and Fellow Eyes) | 645
Primary and Fellow Eyes | 0

6. Other Pre Specified Outcome: Safety Parameter Point Estimate -- (IOP Increase > 10 mmHg) or (IOP > 25 mmHg)
Description: All primary and fellow eyes implanted with the PSI were included in the safety analysis (i.e. both primary and fellow eyes). Point estimates were calculated for the incidence of (IOP Increase > 10 mmHg) or (IOP > 25 mmHg) at the end of the study. Incidence of adverse event totals should not to exceed 5%, and the incidence of each event should not exceed 1-2%.
  NOTE: Because the secondary outcome is a safety measure, both primary and fellow eyes were used for analysis.
Time Frame: as for outcome 2
Population: All subject eyes implanted with the PSI were included in the safety analysis.
Measure: Count of Units; unit: Primary and Fellow Eyes
Units Other Than Participants: Primary and Fellow Eyes
Arm/Group | Overall Study Population
Number analyzed (Participants) | 330
Number analyzed (Primary and Fellow Eyes) | 645
Primary and Fellow Eyes | 55

7. Other Pre Specified Outcome: Safety Parameter Point Estimate -- Chronic Inflammation
Description: All primary and fellow eyes implanted with the PSI were included in the safety analysis. Point estimates were calculated for the incidence of Chronic Inflammation at the end of the study. Incidence of adverse event totals should not to exceed 5%, and the incidence of each event should not exceed 1-2%.
  NOTE: Because the secondary outcome is a safety measure, both primary and fellow eyes were used for analysis.
Time Frame: as for outcome 2
Population: All subject eyes implanted with the PSI were included in the safety analysis.
Measure: Count of Units; unit: Primary and Fellow Eyes
Units Other Than Participants: Primary and Fellow Eyes
Arm/Group | Overall Study Population
Number analyzed (Participants) | 330
Number analyzed (Primary and Fellow Eyes) | 645
Primary and Fellow Eyes | 4

8. Other Pre Specified Outcome: Safety Parameter Point Estimate -- (Axial Length Increase >= 0.20) AND (Myopic Shift > 0.50D MRSE)
Description: All primary and fellow eyes implanted with the PSI were included in the safety analysis. Point estimates were calculated for the incidence of (Axial Length Increase >= 0.20) AND (Myopic Shift > 0.50D MRSE) at the end of the study. Incidence of adverse event totals should not to exceed 5%, and the incidence of each event should not exceed 1-2%.
  NOTE: Because the secondary outcome is a safety measure, both primary and fellow eyes were used for analysis.
Time Frame: as for outcome 2
Population: All subject eyes implanted with the PSI were included in the safety analysis.
Measure: Count of Units; unit: Primary and Fellow Eyes
Units Other Than Participants: Primary and Fellow Eyes
Arm/Group | Overall Study Population
Number analyzed (Participants) | 330
Number analyzed (Primary and Fellow Eyes) | 645
Primary and Fellow Eyes | 0

ADVERSE EVENTS:
Time Frame: Adverse event reporting continued through 24 months.
Groups:
- PresVIEW Implantation - Single Arm: 330 nonrandomized subjects entered into a single group arm to receive the PresView Scleral Implants, which were surgical placed in the sclera of the eye. Subjects were followed for 24 months.
Arm/Group | PresVIEW Implantation - Single Arm
Serious Adverse Events (participants affected / at risk) | 3/330
Other Adverse Events (participants affected / at risk) | 143/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PresVIEW Implantation - Single Arm (N=330)
Decreased iris perfusion (Eye disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PresVIEW Implantation - Single Arm (N=330)
Anterior Eye Structural Change, Deposit and Degeneration (Eye disorders) | 21
Eye Disorders NEC (Eye disorders) | 47
Ocular Hemorrhages and Vascular Disorders NEC (Eye disorders) | 11
Ocular Infections, Irritations and Inflammations (Eye disorders) | 70
Ocular Neoplasms (Eye disorders) | 7
Ocular Neuromuscular Disorders (Eye disorders) | 4
Ocular Sensory Symptoms NEC (Eye disorders) | 8
Ocular Structural Change, Deposit and Degeneration NEC (Eye disorders) | 9
Retina, Choroid and Vitreous Hemorrhages and Vascular Disorders (Eye disorders) | 5
Vision Disorders (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

The Sponsor encourages publication and presentation of the safety and efficacy results upon completion of the study. Per the established agreement, the Principal Investigators will work with the Sponsor, in good faith, to ensure all confidential and proprietary information is redacted.